CLINICAL TRIAL: NCT02011893
Title: Success Using Neuromodulation With BURST (SUNBURST™) Study
Brief Title: SUNBURST (Success Using Neuromodulation With BURST) Study
Acronym: SUNBURST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C-12-07
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Burst Stimulation (Experimental): Burst Stimulation using the Prodigy system
  Interventions: Device: Burst Stimulation
- Tonic Stimulation (Active Comparator): Tonic Stimulation using the Prodigy system
  Interventions: Device: Tonic Stimulation

INTERVENTIONS:
Device: Tonic Stimulation — Prodigy Neurostimulation System with associated components
  Arms: Tonic Stimulation
Device: Burst Stimulation — Prodigy Neurostimulation System with associated components
  Arms: Burst Stimulation

SUMMARY:
The purpose of the study is to demonstrate the safety and efficacy of the Prodigy system for the treatment of chronic intractable pain of the trunk and/or limbs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 22 years of age or older
* Subject has chronic intractable pain of the trunk and/or limbs
* Subject has a average score of 60 or higher for average daily overall pain on the Visual Analog Scale (VAS) 7 day pain diary
* Subject has attempted "best" medical therapy and has tried and failed at least three documented medically supervised treatments (including, but not limited to physical therapy, acupuncture, etc.) and has failed medication treatment from at least two different classes
* Subject's pain-related medication regimen is stable 4 weeks prior to the baseline evaluation
* Subject agrees not to add or increase pain-related medication from activation through the 24 week follow-up visit

Exclusion Criteria:

* Subject is currently participating in a clinical investigation that includes an active treatment arm
* Subject has been implanted with a previous neurostimulation system or participated in a trial period for a neurostimulation system
* Subject's overall Beck Depression Inventory II Score is >24 or has a score of 3 on question 9 relating to suicidal thoughts or wishes at the screening visit
* Subject has an infusion pump or any implantable neurostimulator device
* Subjects with concurrent clinically significant or disabling chronic pain problem that requires additional treatment
* Subject has an existing medical condition that is likely to require repetitive Magnetic Resonance Imaging (MRI) evaluation in the future (i.e. epilepsy, stroke, multiple sclerosis, acoustic neuroma, tumor)
* Subject has an existing medical condition that is likely to require the use of diathermy in the future
* Subject's pain originates from peripheral vascular disease
* Subject is immunocompromised
* Subject has documented history of allergic response to titanium or silicone
* Subject has a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency in the 6 months prior to baseline data collection
* Female candidates of child bearing potential that are pregnant (confirmed by positive urine/blood pregnancy test)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Deer, MD, Study Chair — The Center for Pain Relief
Locations (20):
- United States (20):
  - Newport Beach Headache and Pain, Mission Viejo, California
  - Napa Biomedical Services, Napa, California
  - Eisenhower Desert Orthopedic Center, Rancho Mirage, California
  - IPM Medical Group, Walnut Creek, California
  - Goodman Campbell Brain and Spine, Indianapolis, Indiana
  - Bronson Neuroscience Center, Kalamazoo, Michigan
  - The Neuroscience Center, Biloxi, Mississippi
  - Jackson Pain Center, Jackson, Mississippi
  - Comprehensive Pain & Rehabilitation, Pascagoula, Mississippi
  - Midwest Neurosurgery Associates, Kansas City, Missouri
  - The Montana Center for Wellness & Pain Management, Kalispell, Montana
  - Albany Medical Center, Albany, New York
  - New York Spine & Wellness Center, North Syracuse, New York
  - Oklahoma Pain Physicians, Oklahoma City, Oklahoma
  - NeuroSpine Institute, Eugene, Oregon
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Clinical Trials of South Carolina, North Charleston, South Carolina
  - Houston Pain Centers, Houston, Texas
  - Utah Spine Care, Ogden, Utah
  - The Center for Pain Relief, Charleston, West Virginia

REFERENCES:
- [Derived] Slavin KV, North RB, Deer TR, Staats P, Davis K, Diaz R. Tonic and burst spinal cord stimulation waveforms for the treatment of chronic, intractable pain: study protocol for a randomized controlled trial. Trials. 2016 Dec 1;17(1):569. doi: 10.1186/s13063-016-1706-5. PMID 27906080

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled: All subjects enrolled through device activation/randomization
- Arm 1: Tonic stimulation first, then Burst
- Arm 2: Burst stimulation first, then Tonic
Period: Enrollment to Randomization
Arm/Group | Enrolled | Arm 1 | Arm 2
Started | 173 | 0 | 0
Baseline | 141 | 0 | 0
Trial Stimulation Implant | 121 | 0 | 0
Permanent Stimulation Implant | 101 | 0 | 0
Randomization | 100 | 0 | 0
Completed | 100 | 0 | 0
Not Completed | 73 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Physician Decision | 10 | 0 | 0
Not completed — Withdrawal by Subject | 21 | 0 | 0
Not completed — Screening Failure | 29 | 0 | 0
Not completed — Temporary Trial Stimulation Failure | 9 | 0 | 0
Not completed — Insurance/Financial Reasons | 2 | 0 | 0
Period: Period 1 (Randomization to 12 Weeks)
Arm/Group | Enrolled | Arm 1 | Arm 2
Started | 0 | 45 | 55
6 Week Follow-up | 0 | 45 | 52
12 Week Follow-up | 0 | 45 | 52
Completed | 0 | 45 | 52
Not Completed | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Period: Period 2 (12 Weeks to 24 Weeks)
Arm/Group | Enrolled | Arm 1 | Arm 2
Started | 0 | 45 | 52
18 Week Follow-up | 0 | 44 | 51
24 Week Follow-up | 0 | 45 | 51
Completed | 0 | 45 | 51
Not Completed | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects who were enrolled in the SUNBURST clinical study
Arm/Group | All Subjects
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 56

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Diary Scores for Average Overall Pain
Description: Differences for average daily overall pain using the Visual Analog Scale (VAS) pain diary between Burst and Tonic Stimulation. Visual Analog Scale (VAS) scores were averaged using a 7 day diary where the subject rates his/her pain on a horizontal line, from 0 mm to 100mm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher level of pain.
Time Frame: Over 7 days after 3 months of treatment of burst or tonic stimulation
Population: All subjects randomized were analyzed for this outcome measure. Statistical measures were used to impute Visual Analog Scale (VAS) scores according the study Statistical Analysis Plan (SAP) if data was not available.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Burst Stimulation | Tonic Stimulation
Number analyzed (Participants) | 100 | 100
mm | 43.5 (25.6) | 48.7 (23.9)
Statistical Analysis 1: Comparison: Burst Stimulation vs Tonic Stimulation; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 7.5 points, where the Visual Analog Scale (VAS) scores were measured on a scale of 0 to 100. Testing was carried out at a 5% significance level; p < 0.001, t-distribution; 95% UCB and p-value for non-inferiority are based on t-distribution with n1 + n2-2 degrees of freedom where n1 and n2 are number of subjects per arm

2. Secondary Outcome: Number of Subjects With Response as Measured by Overall Daily Visual Analog Scale (VAS)
Description: Number of subjects responding to Burst and Tonic Stimulation defined as 30% or greater decrease in overall Visual Analog Scale (VAS) score from baseline. Visual Analog Scale (VAS) scores were averaged using a 7 day diary where the subject rates his/her pain on a horizontal line, 100mm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher level of pain.
Time Frame: Over 7 days at baseline and after 3 months of treatment of burst or tonic stimulation
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Burst Stimulation | Tonic Stimulation
Number analyzed (Participants) | 100 | 100
participants | 60 | 51
Statistical Analysis 1: Comparison: Burst Stimulation vs Tonic Stimulation; Test type: Superiority or Other; p = 0.083, McNemar — Superiority analysis performed

3. Secondary Outcome: Percentage of Paresthesia Coverage
Description: Paresthesia mapping (percentage of paresthesia coverage) analyzed to demonstrate the differences between Burst and Tonic Stimulation. Data is presented as areas of paresthesia reported while utilizing either Burst or Tonic Stimulation as a percentage of the total number of areas possible.
Time Frame: During in-office visit after 3 months of treatment while utilizing burst or tonic stimulation
Population: There were 73 subjects in whom paresthesia coverage data at both the 12 and 24 week visits were available and included in the analysis. The remaining 23 subjects were excluded due to questionnaire completion errors at the time of data collection.
Measure: Mean (Standard Deviation); unit: Percentage of paresthesia areas
Arm/Group | Burst Stimulation | Tonic Stimulation
Number analyzed (Participants) | 73 | 73
Percentage of paresthesia areas | 4.5 (8.7) | 22.7 (16.3)

4. Secondary Outcome: Test for Superiority of Overall Daily Visual Analog Scale (VAS) Score With Burst Stimulation
Description: Differences for average daily overall pain using the Visual Analog Scale (VAS) pain diary between Burst and Tonic Stimulation to evaluate for superiority of Burst Stimulation. Differences for average daily overall pain using the Visual Analog Scale (VAS) pain diary between Burst and Tonic Stimulation. Visual Analog Scale (VAS) scores were averaged using a 7 day diary where the subject rates his/her pain on a horizontal line, 100mm in length, anchored by word descriptors on each end (no pain to worst imaginable pain). A higher score indicates a higher level of pain.
Time Frame: Over 7 days after 3 months of treatment of burst or tonic stimulation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Burst Stimulation | Tonic Stimulation
Number analyzed (Participants) | 100 | 100
mm | 43.5 (25.6) | 48.7 (23.9)
Statistical Analysis 1: Comparison: Burst Stimulation vs Tonic Stimulation; Test type: Superiority or Other; p = 0.017, t-distribution — Superiority analysis performed; 95% UCB and p-value for superiority are based on t-distribution with n1 + n2-2 degrees of freedom where n1 and n2 are number of subjects per arm

ADVERSE EVENTS:
Time Frame: following enrollment through 6 months of treatment
Description: Subjects at risk (denominators for risk %) are defined as follows: enrollment to device activation (randomization) is 173, device activation (randomization) to 24 weeks is 100. The only events identified as device (stimulation) related are reported per intervention, by therapy (Burst and Tonic Stimulation). The subjects at risk (denominators for risk %) for are defined as follows: subjects active through 12 weeks (100) or subjects active through 24 weeks (97).
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 12/173
Other Adverse Events (participants affected / at risk) | 13/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | All Subjects (N=173)
Persistent pain and/or numbness (Injury, poisoning and procedural complications) | 1 (1) — Categorized as Procedure-Related
Unsuccessful lead placement (Injury, poisoning and procedural complications) | 1 (1) — Categorized as Procedure-Related
Abdominal pain (Hepatobiliary disorders) | 1 (1) — Categorized as neither Device- nor Procedure-Related
Bowel obstruction (Gastrointestinal disorders) | 1 (1) — Categorized as neither Device- nor Procedure-Related
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) — Categorized as neither Device- nor Procedure-Related
Hip pain/hip replacement (Surgical and medical procedures) | 1 (1) — Categorized as neither Device- nor Procedure-Related
Low Potassium Levels (General disorders) | 1 (1) — Categorized as neither Device- nor Procedure-Related
Persistent pain and/or numbness (Injury, poisoning and procedural complications) | 1 (1) — Categorized as neither Device- nor Procedure-Related
Cancerous tumor on vocal chords (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/100 (1) — Categorized as neither Device- nor Procedure-Related
Infection (Infections and infestations) | 1/100 (1) — Categorized as neither Device- nor Procedure-Related
Loss of speech and memory, and headache (Nervous system disorders) | 1/100 (1) — Categorized as neither Device- nor Procedure-Related
Scheduled right total knee arthroplasty (Surgical and medical procedures) | 1/100 (1) — Categorized as neither Device- nor Procedure-Related
Shortness of breath (Cardiac disorders) | 1/100 (1) — Categorized as neither Device- nor Procedure-Related
Somnolence (General disorders) | 1/100 (1) — Categorized as neither Device- nor Procedure-Related
Temporary paralysis (Nervous system disorders) | 1/100 (1) — Categorized as neither Device- nor Procedure-Related
Withdrawal symptoms from tapering off oxymorphone (General disorders) | 1/100 (1) — Categorized as neither Device- nor Procedure-Related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | All Subjects (N=100)
Diminished or loss of symptom relief (Burst Stimulation) (General disorders) | 5 (5) — Categorized as Device-Related
Diminished or loss of symptom relief (Tonic Stimulation) (General disorders) | 6/97 (8) — Categorized as Device-Related
Persistent pain and/or numbness (General disorders) | 8 (8) — Categorized as neither Device- nor Procedure-Related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other